CLINICAL TRIAL: NCT02691078
Title: Validation of 99mTc- EDDA - HYNIC -TOC Kits for Diagnosis of Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Financiadora de Estudos e Projetos (Other); Instituto do Cérebro do Rio Grande do Sul - InsCer (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LACOG 0214
Record Dates: First submitted 2016-02-11; First posted 2016-02-25 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adult patients with neuroendocrine tumors (Experimental)
  Interventions: Other: 99m Tc - HYNIC -TOC EDDA and 111In - DTPA-octreotide

INTERVENTIONS:
Other: 99m Tc - HYNIC -TOC EDDA and 111In - DTPA-octreotide — The patient will undercome an PET/CT exam with 99m Tc - HYNIC -TOC EDDA, after 20 days of wash out, the same patient will undercome the same exam with 111In - DTPA-octreotide in order to compare both radiopharmaceuticals

SUMMARY:
Evaluation of the properties of the image capture test using 99m Tc - HYNIC -TOC EDDA (octreotide labeled with 99mTc) for the diagnosis of neuroendocrine tumors compared to the 111In - DTPA-octreotide.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of neuroendocrine tumors
* Patients with indication for the staging exam with 11In
* Patients diagnosed in any tumor stage
* Patients with > 18 years
* Male and female patients
* Patients not receiving somatostatin analogues for at least 1 month before image capturing

Exclusion Criteria:

* Pregnant women
* Patients with previous tumor resection of the primary tumor without metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Analysis of the images captured with 99m Tc - HYNIC -TOC EDDA ( octreotide labeled with 99mTc ) and 111In - DTPA-octreotide for the diagnosis of neurocrine tumors | Up to 30 days

SECONDARY OUTCOMES:
Visualization of the ocurrence of the neuroendocrine tumor lesions with both radiopharmaceutical agents | Up to 30 days
Number of neuroendocrine tumor lesions visualized with both radiopharmaceutical agents | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group
Locations (1):
- Instituto do Cérebro do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Moriguchi-Jeckel CM, Madke RR, Radaelli G, Viana A, Nabinger P, Fernandes B, Gossling G, Berdichevski EH, Vilas E, Giacomazzi J, Rocha MS, Borges JA, Hoffmann E, Greggio S, Venturin GT, Barrios CH, Zaffaroni F, Werutsky G, da Costa JC. Clinical validation and diagnostic accuracy of 99mTc-EDDA/HYNIC-TOC compared to 111In-DTPA-octreotide in patients with neuroendocrine tumours: the LACOG 0214 study. Ecancermedicalscience. 2023 Jul 26;17:1582. doi: 10.3332/ecancer.2023.1582. eCollection 2023. PMID 37533941
- See also: Disclosure of the study on the sponsor's website. — http://lacogcancerresearch.org/studies/clinical-trials/closed/lacog-0214-finep/